CLINICAL TRIAL: NCT00027170
Title: Technical Development of Cardiovascular Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020050; 02-H-0050
Record Dates: First submitted 2001-11-27; First posted 2001-11-28 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2020-12-22

CONDITIONS: Cardiomyopathy; Congenital Heart Disease; Cardiovascular Disease; Cardiac Magnetic Resonance Imaging; Acute Myocardial Infarction
Keywords: Myocardial Infarction; Myocardial Viability; Myocardial Perfusion; Myocardial Ischemia; Atherosclerosis
MeSH Terms: conditions — Cardiomyopathies; Heart Defects, Congenital; Cardiovascular Diseases; Myocardial Infarction; Myocardial Ischemia; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Participants with cardiovascular diseases: Patients may receive an intravenous injection of gadobutrol (Gadavist) not to exceed 0.2 mmol/kg of Gd per bolus injection and per examination.
  Interventions: Device: Siemens MRI scanner
- Healthy Participants: Patients may receive an intravenous injection of gadobutrol (Gadavist) not to exceed 0.2 mmol/kg of Gd per bolus injection and per examination.
  Interventions: Device: Siemens MRI scanner

INTERVENTIONS:
Device: Siemens MRI scanner — Investigational or research MRI coils may be used in the protocol. The coils are noninvasive devices external to the body. The coils act as antennae to receive small radiofrequency signals out of the body. Coils of the type we use are used daily in clinical MRI practice.

SUMMARY:
This study will explore new ways of using magnetic resonance imaging (MRI) to evaluate the heart and blood vessels of patients with cardiovascular disease, including better detection of myocardial infarction (heart attack) and blockage of heart and leg arteries.

Patients 18 years of age and older with cardiovascular disease may be eligible for this study.

All participants will have magnetic resonance imaging of the heart. MRI uses a magnetic field and radio waves to show structural and chemical changes in tissues. For the procedure, the patient lies on a table surrounded by a metal cylinder (the scanner). A 'gadolinium contrast' material may be injected into the patient s vein during part of the study to brighten the images. Patients wear earplugs during the scan to muffle loud knocking sounds caused by the electrical switching of the magnetic fields. They will be asked to hold their breath intermittently for 5 to 20 seconds during the scan. They will be monitored with an electrocardiogram (EKG) during the procedure and will be in contact by intercom at all times with the person performing the scan. Patients can request to stop the study and come out of the scanner at any time. The procedure may last from 30 to 90 minutes. An echocardiogram a test that uses sound waves to produce pictures of the heart and blood vessels-may be done to confirm the MRI findings. In addition, patients may undergo one or more of the following optional studies:

* Dobutamine stress MRI - This test uses dobutamine-a medicine that simulates exercise by increasing heart rate and heart function-to detect blockages in the coronary arteries (vessels that supply oxygen and nutrients to the heart) and locate areas of the heart that are permanently damaged, perhaps by a previous heart attack. For this test, MRI pictures of the heart are taken before, during and after administration of dobutamine. Gadolinium may be injected during part of the study to brighten the images. An EKG will be used to monitor the heart during the procedure.
* Vasodilator MRI - The procedure and objectives of this test are the same as those described for dobutamine stress MRI, except that this study uses dipyridamole or adenosine. These drugs dilate blood vessels, causing increased blood flow to the heart.
* Plethysmography MRI - This test determines the presence and severity of narrowing in arteries that supply blood to the leg. Blockage of these vessels often causes pain while walking. This study will compare plethysmography MRI with venous occlusion plethysmography, an older method of measuring blood flow in the legs. For venous occlusion plethysmography, a large blood pressure cuff is placed around the upper leg and a strain gauge (thin elastic band) is placed around the calf. The pressure cuff is inflated very tightly for 5 minutes to block blood flow to the leg, and another pressure cuff over the ankle is also inflated. When the large cuff is deflated, blood rushes to the leg, a smaller cuff is inflated to a low pressure, and the strain gauge measures the maximum blood flow to the leg for 1 or 2 more minutes. This procedure is done once or twice outside the MRI scanner and once or twice inside the scanner. The scans are performed as described above for the dobutamine and vasodilator studies. The strain gauge is not used for plethysmography MRI the MRI pictures are used to measure flow.

DETAILED DESCRIPTION:
The purpose of this protocol is to allow development and testing of new MRI techniques suitable for evaluating patients with cardiovascular disease. Since such technical development work often depends on preliminary studies in healthy volunteers, the protocol also recruits healthy subjects. This protocol will provide the framework for technical development scans in patients with cardiovascular disease.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Inclusion Criteria for All Arms of the Protocol:

   * Subjects 18 years of age or older
   * Written informed consent

   EXCLUSION CRITERIA:
2. Exclusion Criteria for All Arms of the Protocol:

   * Patients with a contraindication to MRI scanning will be excluded. These contraindications include patients with the following devices:

     * Central nervous system aneurysm clips;
     * Implanted neural stimulator;
     * Implanted cardiac pacemaker or defibrillator;
     * Cochlear implant;
     * Ocular foreign body (e.g. metal shavings);
     * Implanted Insulin pump;
     * Metal shrapnel or bullet.
3. In addition, the following patient groups will be excluded:

   * Pregnant women (Patients who are uncertain as to whether they are pregnant will be required to have a screening urine or blood pregnancy test)
   * Patients with active symptoms of myocardial ischemia occurring despite maximally tolerated doses of oral antianginal therapy and intravenous nitroglycerin
4. Furthermore, the following patient groups will be excluded from studies involving the administration of MRI contrast agents:

   * lactating women unless they are willing to discard breast milk for 24 hours after receiving gadolinium
   * renal disease (estimated glomerular filtration rate (eGFR) less than 30 ml/min/1.73 m(2) body surface area)

   The eGFR will be used to estimate renal function if reported by the laboratory, or as reported by NIH Clinical Center or Suburban Hospital or other clinically certified laboratories. Otherwise, estimated glomerular filtration rate (eGFR) can be based on the Modification of Diet in Renal Disease (MDRD) study equation (see below) in subjects with stable renal function. This formula is not applicable to patients with acute renal insufficiency:

   eGFR (ml/min/1.73 m(2)) equal to 175 times (serum creatinine)-1.154 times (age)-0.203 times 0.742 (if the subject is female) times1.212 (if the subject is black)
5. Additional Exclusion Criteria for Dobutamine, or Vasodilator Stress MRI:

   * Myocardial infarction within 48 hours
   * Uncontrolled congestive heart failure
   * Severe hypertension (SBP greater than 200, DBP greater than 110) (exclusion only for dobutamine and bicycle)
   * Atrial fibrillation. This exclusion only applies to Dobutamine stress.
   * Frequent PVC s (more than 1 every 10 heart beats or non-sustained ventricular tachycardia (greater than 4 beat runs) or ongoing sustained ventricular tachycardia. This exclusion only applies to Dobutamine and Bicycle stress
   * Patients with narrow angle glaucoma and known or suspected prostatic obstruction will not receive atropine
6. Additional Exclusion Criteria for PET/MR perfusion scans

   * Pregnant patients
   * Patients that are breast feeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiovascular diseases and healthy subjects 18 years of age or older were recruited within this protocol. The exclusion criteria were developed from standard clinical practice but were more restrictive to err on the side of safety. Recruitment was via referral from local physicians. In addition, advertisements were placed in the "Washington Post". Finally, the protocol was listed on the NIH websites.
  A patient could participate in any combination of these tests/procedures. Clinical judgment was used to determine the number of tests/procedures suitable for a given patient. Specifically, the responsible physician avoided prolonging tests/procedures in patients in accordance with the patient's clinical status.
Sampling Method: Non-Probability Sample
Enrollment: 8781 (Actual)
Dates: Start 2001-11-26 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
examine the rate of major cardiovascular events (MACE) defined as cardiac death, non- fatal myocardial infarction, cerebrovascular / transient ischemic attack, and revascularization in patients undergoing stress or rest cardiac MRI | Ongoing
  examine the rate of major cardiovascular events (MACE) defined as cardiac death, non- fatal myocardial infarction, cerebrovascular / transient ischemic attack, and revascularization in patients undergoing stress or rest cardiac MRI and to relate these events to the extent of ischemia and infarction seen on the MRI exams

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Sirajuddin, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Baer FM, Voth E, Theissen P, Schicha H, Sechtem U. Gradient-echo magnetic resonance imaging during incremental dobutamine infusion for the localization of coronary artery stenoses. Eur Heart J. 1994 Feb;15(2):218-25. doi: 10.1093/oxfordjournals.eurheartj.a060479. PMID 8005123
- [Background] Baer FM, Voth E, Schneider CA, Theissen P, Schicha H, Sechtem U. Comparison of low-dose dobutamine-gradient-echo magnetic resonance imaging and positron emission tomography with [18F]fluorodeoxyglucose in patients with chronic coronary artery disease. A functional and morphological approach to the detection of residual myocardial viability. Circulation. 1995 Feb 15;91(4):1006-15. doi: 10.1161/01.cir.91.4.1006. PMID 7850935
- [Background] Baer FM, Voth E, Theissen P, Schneider CA, Schicha H, Sechtem U. Coronary artery disease: findings with GRE MR imaging and Tc-99m-methoxyisobutyl-isonitrile SPECT during simultaneous dobutamine stress. Radiology. 1994 Oct;193(1):203-9. doi: 10.1148/radiology.193.1.8090892.
- [Derived] Fujikura K, Sathya B, Acharya T, Benovoy M, Jacobs M, Sachdev V, Hsu LY, Arai AE. CMR provides comparable measurements of diastolic function as echocardiography. Sci Rep. 2024 May 22;14(1):11658. doi: 10.1038/s41598-024-61992-6. PMID 38778036
- [Derived] Ta AD, Hsu LY, Conn HM, Winkler S, Greve AM, Shanbhag SM, Chen MY, Patricia Bandettini W, Arai AE. Fully quantitative pixel-wise analysis of cardiovascular magnetic resonance perfusion improves discrimination of dark rim artifact from perfusion defects associated with epicardial coronary stenosis. J Cardiovasc Magn Reson. 2018 Mar 8;20(1):16. doi: 10.1186/s12968-018-0436-0. PMID 29514708
- [Derived] Hsu LY, Jacobs M, Benovoy M, Ta AD, Conn HM, Winkler S, Greve AM, Chen MY, Shanbhag SM, Bandettini WP, Arai AE. Diagnostic Performance of Fully Automated Pixel-Wise Quantitative Myocardial Perfusion Imaging by Cardiovascular Magnetic Resonance. JACC Cardiovasc Imaging. 2018 May;11(5):697-707. doi: 10.1016/j.jcmg.2018.01.005. Epub 2018 Feb 14. PMID 29454767
- [Derived] Nielles-Vallespin S, Kellman P, Hsu LY, Arai AE. FLASH proton density imaging for improved surface coil intensity correction in quantitative and semi-quantitative SSFP perfusion cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2015 Feb 17;17(1):16. doi: 10.1186/s12968-015-0120-6. PMID 25827180
- [Derived] Chen MY, Bandettini WP, Shanbhag SM, Vasu S, Booker OJ, Leung SW, Wilson JR, Kellman P, Hsu LY, Lederman RJ, Arai AE. Concordance and diagnostic accuracy of vasodilator stress cardiac MRI and 320-detector row coronary CTA. Int J Cardiovasc Imaging. 2014 Jan;30(1):109-19. doi: 10.1007/s10554-013-0300-0. Epub 2013 Oct 12. PMID 24122452
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-H-0050.html